CLINICAL TRIAL: NCT06406712
Title: Efficacy of Retroclavicular Dexamethasone With Bupivacaine in Patients Undergoing Upper Limb Vascular Surgeries
Brief Title: Retroclavicular Block in Vascular Surgey
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Abdelsabour, lecture of anesthesia and ICU, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: new valley anesthesia g2
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone with bupivacaine in retroclavicular block (Active Comparator): 40patients received 40 ml of bupivacaine 0.25%(in total 100 mg)+1 ml of dexamethasone)
  Interventions: Other: retroclavicular block
- bupivacaine in retroclavicular block (control group) (Active Comparator): : 40patients received. 40 ml of bupivacaine 0.25%(in total 100 mg)+1 ml saline
  Interventions: Other: retroclavicular block

INTERVENTIONS:
Other: retroclavicular block — regional anesthesia

SUMMARY:
The retroclavicular (coracoid) approach for brachial plexus anesthesia is recognized for its facility and simplicity to perform .

The block has been well described in the anesthesia community since it was first introduced by Hebbard and Royse in 2007 . In 2017, Luftig . first described the block's use in the ED setting for a variety of indications . Because of its different needle entry point, the retro clavicular (RCB) approach offers an almost perpendicular needle-ultrasound (US) beam angle.

DETAILED DESCRIPTION:
Regional anesthesia (RA) offers several advantages over general anesthesia (GA) for upper limb orthopedic surgery. One of the advantages is the improvement in postoperative pain, which leads to decreased use of postoperative opioids needs and reduces the recovery time for patients . A variety of approaches for regional blockade for upper extremity surgery have been described.

Dexamethasone is a corticosteroid drug that has been used as an adjuvant to reduce postoperative pain.

The use of peri neural dexamethasone (i.e. dexamethasone added to the local anesthesia solution) as an adjuvant to peripheral nerve block to improve analgesia provided by local anesthetic alone . Peri neural dexamethasone, as an adjuvant to peripheral nerve block, has been associated with faster onset of anesthesia , longer duration of anesthesia/analgesia decreased postoperative pain intensity and decreased postoperative analgesia requirements compared with local anaesthetic alone . The exact mechanism by which dexamethasone reduces pain is not known. The decrease in pain intensity and the prolonged analgesia attained with the use of perineural dexamethasone may be the result of a local, or systemic action, or both . Dexamethasone may act locally on glucocorticosteroid receptors to induce vasoconstriction, thereby decreasing systemic absorption of local anaesthetics . Other potential mechanisms of action include suppression of C-fibre transmission of pain signals and direct action on the nerve cell to reduce neural discharge . Dexamethasone may act systemically by reducing the inflammatory response caused by surgical tissue injury .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper limb vascular surgey .

Exclusion Criteria:

* - Contraindications to regional block (coagulopathy, infection at the needle insertion site, or diaphragmatic paralysis).
* Altered conscious level.
* Pregnancy.
* Body mass index (BMI > 35).
* Patients who have difficulty understanding the study protocol.
* Patients who have any known contraindication to study medications.
* Patient refusal.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
sensory and motor duration of block | 24 hours
  efficacy of block

CONTACTS AND LOCATIONS:
Overall Officials: ahmed ismail, lecture, Principal Investigator — faculty of medicine , new valley university
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No